CLINICAL TRIAL: NCT06594757
Title: Evaluation of Plaque Removal by Triple-Headed Manual Toothbrush: A Randomized Controlled Clinical Trial
Brief Title: Plaque Removal by Triple-Headed Manual Toothbrush
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Didem OZKAL EMINOGLU, Assistant Professor, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: TSA-2023-13318
Record Dates: First submitted 2024-09-09; First posted 2024-09-19 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Plaque, Dental
Keywords: oral hygiene; Rustogi Modifiye Navy Plaque Index; Modified Bass Technique; toothbrush; dental plaque
MeSH Terms: conditions — Dental Plaque | interventions — Toothbrushing

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standart Manual Toothbrush (SMB) (Active Comparator): Conventional toothbrushing with standart manual toothbrush
  Interventions: Procedure: Toothbrushing with standard manual toothbrush
- Triple-Headed Manual Toothbrush (3HB) (Experimental): Toothbrushing with triple-headed manual toothbrush
  Interventions: Procedure: Toothbrushing with triple-headed manual toothbrush

INTERVENTIONS:
Procedure: Toothbrushing with triple-headed manual toothbrush — Toothbrushing with triple-headed manual toothbrush
  Arms: Triple-Headed Manual Toothbrush (3HB)
Procedure: Toothbrushing with standard manual toothbrush — Toothbrushing with tstandard manual toothbrush
  Arms: Standart Manual Toothbrush (SMB)

SUMMARY:
This randomized controlled trial aimed to determine the effectiveness of a plaque removal by triple-headed manual toothbrush by comparing changes in Rustogi Modifiye Navy Plaque Index.

Participants will be divided into two groups and will be made to brush with different designed toothbrushes.

The researchers will compare the plaque removal efficiency of the brushes by comparing the changes in the plaque index of the intervention and control groups before and after brushing.

ELIGIBILITY:
Inclusion Criteria:

* age ranging from 18-60 years;
* a minimum of 12 teeth;
* participants were wanted to be right-handers when toothbrushing to standardization.

Exclusion Criteria:

* Patients with systemic illnesses or conditions,
* smokers and individuals taking any medication that may affect periodontal health were not included in the study.
* Individuals who had previously been treated for periodontal disease in the past 6 months were also excluded.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Rustogi Modifiye Navy Plaque Index | 1 minute before brushing
  The amount of plaque present on the teeth was assessed using a plaque staining agent and graded according to the plaque index system. Higher scores mean a worse outcome.
Rustogi Modifiye Navy Plaque Index | 1 minute after brushing
  The amount of plaque present on the teeth was assessed using a plaque staining agent and graded according to the plaque index system. Higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Didem Özkal Eminoğlu, Study Director — Ataturk University
Locations (1):
- Atatürk University, Erzurum, Turkey (Türkiye)